CLINICAL TRIAL: NCT03022396
Title: Protective Mechanisms Against a Pandemic Respiratory Virus: B- Cell, T-cell, and General Immune Response to Seasonal Influenza Vaccine. Year 2, 2010
Brief Title: T-cell And General Immune Response to Seasonal Influenza Vaccine (SLVP018) Year 2, 2010
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Cornelia L. Dekker, Professor, Pediatrics, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SU-17219-2010; 2U19AI057229-06 (NIH)
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Results first posted 2017-08-21 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Influenza
Keywords: Inactivated influenza vaccine; Identical twins; Fraternal twins; High-Dose influenza vaccine; Elderly twins; Child twins; Inactivated influenza vaccine, high-dose
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Injections, Intramuscular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group A: age 8-17 yo identical twins (Other): Individual twins to receive Fluzone® (intramuscular)
  Interventions: Biological: Fluzone® (intramuscular)
- Group B: age 18-30 yo identical twins (Other): Individual twins to receive Fluzone® (intramuscular)
  Interventions: Biological: Fluzone® (intramuscular)
- Group C: age 18-30 yo fraternal twins (Other): Individual twins to receive Fluzone® (intramuscular)
  Interventions: Biological: Fluzone® (intramuscular)
- Group D: age 40 - 59 yo identical twins (Other): Individual twins to receive Fluzone® (intramuscular)
  Interventions: Biological: Fluzone® (intramuscular)
- Group E: age 40 - 59 yo fraternal twins (Other): Individual twins to receive Fluzone® (intramuscular)
  Interventions: Biological: Fluzone® (intramuscular)
- Group F: age 70 - 100 yo identical twins (Other): Individual twins to receive Fluzone® (intramuscular) or High Dose Fluzone® (intramuscular)
  Interventions: Biological: High Dose Fluzone® (intramuscular); Biological: Fluzone® (intramuscular)

INTERVENTIONS:
Biological: High Dose Fluzone® (intramuscular) — Licensed seasonal High dose trivalent inactivated influenza
  Other Names: High Dose TIV
  Arms: Group F: age 70 - 100 yo identical twins
Biological: Fluzone® (intramuscular) — Licensed seasonal trivalent inactivated influenza
  Other Names: TIV

SUMMARY:
This study will investigate response to influenza vaccines in monozygotic and dizygotic twins of different ages.

DETAILED DESCRIPTION:
The investigators plan to study the response to influenza vaccines much more broadly and deeply across different age groups and with different vaccine formulations and to probe the influence of genetics on these responses using monozygotic and dizygotic twins. On an investigational basis, investigators plan to compare various immunological responses, identify age-specific biomarkers or clusters of markers, quantify the frequency of influenza-specific T-cells pre- and post-vaccination, and determine the effective breadth of T-cell repertoire to an influenza vaccine within an individual as a function of age and to what degree this is genetically determined.

Twin Groups A-E will receive a single administration of the 2010-2011 formulation of seasonal trivalent inactivated influenza vaccine (TIV). Group F, elderly monozygotic twin participants, will be randomly assigned to receive a single dose of inactivated vaccine, either the usual dose or the High-Dose TIV. Blood samples to conduct the assays described will be taken at pre-immunization, Days 7-10 and 28 post-immunization. Each twin is counted as a single participant. All reporting numbers reflect the number of participants, not the number of twin pairs.

ELIGIBILITY:
Inclusion Criteria:

1. Otherwise healthy, ambulatory children or adults, ages 8-17 years (identical twins), 18-30 years (identical or fraternal twins), 40-59 years (identical or fraternal twins) or 70-100 years (identical twins).
2. Willing to complete the informed consent process.
3. Availability for follow-up for the planned duration of the study at least 28 days after immunization.
4. Acceptable medical history and vital signs.
5. All female of childbearing potential, must use an acceptable method of contraception and not become pregnant for the duration of the study (approximately 1 month or to completion of Visit 3). (Acceptable contraception includes implants, injectables, combined oral contraceptives, effective intrauterine devices (IUDs), sexual abstinence, or a vasectomized partner).

Exclusion Criteria:

1. Prior off-study vaccination with trivalent inactivated influenza vaccine (TIV) or live attenuated influenza vaccine (LAIV) in Fall 2010
2. Allergy to egg or egg products, or to vaccine components, including thimerosal (if TIV multidose vials used)
3. Life-threatening reactions to previous influenza vaccinations
4. Active systemic or serious concurrent illness, including febrile illness on the day of vaccination
5. History of immunodeficiency
6. Known or suspected impairment of immunologic function, including, but not limited to, clinically significant liver disease, diabetes mellitus treated with insulin, moderate to severe renal disease or any other chronic disorder which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
7. Blood pressure >150 systolic or > 95 diastolic at Visit 1
8. Hospitalization in the past year for congestive heart failure or emphysema.
9. Chronic Hepatitis B or C
10. Recent or current use of immunosuppressive medication, including glucocorticoids (corticosteroid nasal sprays and inhaled steroids are permissible). Use of oral steroids (<20mg prednisone-equivalent/day) may be acceptable after review by the investigator.
11. Malignancy, other than squamous cell or basal cell skin cancer (includes solid tumors such as breast cancer or prostate cancer with recurrence in the past year, and any hematologic cancer such as leukemia).
12. Autoimmune disease (including rheumatoid arthritis treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
13. History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year
14. Use of any anti-coagulation medication such as Coumadin or Lovenox, or anti-platelet agents such as aspirin, Plavix, Aggrenox must be reviewed by investigator to determine if this would affect the volunteer's safety.
15. Receipt of blood or blood products within the past 6 months
16. Medical or psychiatric condition or occupational responsibilities that preclude subject compliance with the protocol
17. Inactivated vaccine 14 days prior to vaccination
18. Live, attenuated vaccine within 60 days of vaccination
19. History of Guillain-Barre Syndrome
20. Pregnant or lactating woman
21. Use of investigational agents within 30 days prior to enrollment
22. Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment
23. Any condition which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol.

Ages: 8 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Dekker, MD, Principal Investigator — Stanford University; Mark Davis, PhD, Principal Investigator — Stanford University; Garry Nolan, PhD, Principal Investigator — Stanford University; Ann Arvin, MD, Principal Investigator — Stanford University; Stephen Quake, PhD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horowitz A, Strauss-Albee DM, Leipold M, Kubo J, Nemat-Gorgani N, Dogan OC, Dekker CL, Mackey S, Maecker H, Swan GE, Davis MM, Norman PJ, Guethlein LA, Desai M, Parham P, Blish CA. Genetic and environmental determinants of human NK cell diversity revealed by mass cytometry. Sci Transl Med. 2013 Oct 23;5(208):208ra145. doi: 10.1126/scitranslmed.3006702. PMID 24154599
- [Background] Kay AW, Fukuyama J, Aziz N, Dekker CL, Mackey S, Swan GE, Davis MM, Holmes S, Blish CA. Enhanced natural killer-cell and T-cell responses to influenza A virus during pregnancy. Proc Natl Acad Sci U S A. 2014 Oct 7;111(40):14506-11. doi: 10.1073/pnas.1416569111. Epub 2014 Sep 22. PMID 25246558
- [Background] Brodin P, Jojic V, Gao T, Bhattacharya S, Angel CJ, Furman D, Shen-Orr S, Dekker CL, Swan GE, Butte AJ, Maecker HT, Davis MM. Variation in the human immune system is largely driven by non-heritable influences. Cell. 2015 Jan 15;160(1-2):37-47. doi: 10.1016/j.cell.2014.12.020. PMID 25594173
- [Background] Kay AW, Bayless NL, Fukuyama J, Aziz N, Dekker CL, Mackey S, Swan GE, Davis MM, Blish CA. Pregnancy Does Not Attenuate the Antibody or Plasmablast Response to Inactivated Influenza Vaccine. J Infect Dis. 2015 Sep 15;212(6):861-70. doi: 10.1093/infdis/jiv138. Epub 2015 Mar 4. PMID 25740957
- [Background] Rubelt F, Bolen CR, McGuire HM, Vander Heiden JA, Gadala-Maria D, Levin M, Euskirchen GM, Mamedov MR, Swan GE, Dekker CL, Cowell LG, Kleinstein SH, Davis MM. Individual heritable differences result in unique cell lymphocyte receptor repertoires of naive and antigen-experienced cells. Nat Commun. 2016 Mar 23;7:11112. doi: 10.1038/ncomms11112. PMID 27005435
- [Background] Horns F, Vollmers C, Croote D, Mackey SF, Swan GE, Dekker CL, Davis MM, Quake SR. Lineage tracing of human B cells reveals the in vivo landscape of human antibody class switching. Elife. 2016 Aug 2;5:e16578. doi: 10.7554/eLife.16578. PMID 27481325
- [Derived] Cheung P, Vallania F, Warsinske HC, Donato M, Schaffert S, Chang SE, Dvorak M, Dekker CL, Davis MM, Utz PJ, Khatri P, Kuo AJ. Single-Cell Chromatin Modification Profiling Reveals Increased Epigenetic Variations with Aging. Cell. 2018 May 31;173(6):1385-1397.e14. doi: 10.1016/j.cell.2018.03.079. Epub 2018 Apr 26. PMID 29706550
- [Derived] de Bourcy CFA, Dekker CL, Davis MM, Nicolls MR, Quake SR. Dynamics of the human antibody repertoire after B cell depletion in systemic sclerosis. Sci Immunol. 2017 Sep 29;2(15):eaan8289. doi: 10.1126/sciimmunol.aan8289. PMID 28963118

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All numbers of participants reflect an individual participant, not a twin pair. All enrollment numbers reflect the number of participants, not the number of twin pairs.
Period: Overall Study
Arm/Group | Group A: Age 8-17 yo Identical Twins | Group B: Age 18-30 yo Identical Twins | Group C: Age 18-30 yo Fraternal Twins | Group D: Age 40 - 59 yo Identical Twins | Group E: Age 40 - 59 yo Fraternal Twins | Group F: Age 70 - 100 yo Identical Twins
Started | 16 | 14 | 10 | 20 | 14 | 8
Completed | 16 | 14 | 10 | 20 | 14 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All numbers reflect the number of individual participants, not the number of twin pairs. Ie, in Group A there were 16 participants who were part of 8 twin pairs.
Groups:
- Group F: Age 70 - 100 yo Twins: Individual twins to receive Fluzone® (intramuscular) or High Dose Fluzone® (intramuscular)
  High Dose Fluzone® (intramuscular): Licensed seasonal High dose trivalent inactivated influenza
  Fluzone® (intramuscular): Licensed seasonal trivalent inactivated influenza
- Total: Total of all reporting groups
Arm/Group | Group A: Age 8-17 yo Identical Twins | Group B: Age 18-30 yo Identical Twins | Group C: Age 18-30 yo Fraternal Twins | Group D: Age 40 - 59 yo Identical Twins | Group E: Age 40 - 59 yo Fraternal Twins | Group F: Age 70 - 100 yo Twins | Total
Number analyzed (Participants) | 16 | 14 | 10 | 20 | 14 | 8 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.69 (1.88) | 23.71 (3.33) | 22.65 (2.99) | 53.44 (2.25) | 44.52 (1.68) | 75.51 (4.50) | 37.70 (19.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 3 | 14 | 13 | 2 | 48
  Male | 8 | 6 | 7 | 6 | 1 | 6 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2 | 2 | 0 | 0 | 6
  Not Hispanic or Latino | 16 | 12 | 8 | 18 | 14 | 8 | 76
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — The Race is inconsistent in Group D because identical twins self reported differently from each other. One identical twin reported Hispanic and American Indian and the other identical twin said Hispanic and Caucasian.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1
    Asian | 0 | 2 | 3 | 0 | 1 | 0 | 6
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 4 | 0 | 4
    White | 10 | 9 | 6 | 19 | 8 | 8 | 60
    More than one race | 6 | 2 | 1 | 0 | 1 | 0 | 10
    Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 14 | 10 | 20 | 14 | 8 | 82

OUTCOME MEASURES:

1. Primary Outcome: Number of Individual Twins Who Received Influenza Vaccine
Description: All numbers reported are the number of participants, not the number of twin pairs. Each member of a twin was counted individually as a participant.
Time Frame: Day 0 to 28
Population: All numbers reported are the number of participants, not the number of twin pairs. Each member of a twin was counted individually as a participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Age 8-17 yo Identical Twins | Group B: Age 18-30 yo Identical Twins | Group C: Age 18-30 yo Fraternal Twins | Group D: Age 40 - 59 yo Identical Twins | Group E: Age 40 - 59 yo Fraternal Twins | Group F: Age 70 - 100 yo Twins
Number analyzed (Participants) | 16 | 14 | 10 | 20 | 14 | 8
Participants | 16 | 14 | 10 | 20 | 14 | 8

2. Secondary Outcome: Number of Individual Twins With Related Adverse Events
Time Frame: Day 0 to 28 post-immunization
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Age 8-17 yo Identical Twins | Group B: Age 18-30 yo Identical Twins | Group C: Age 18-30 yo Fraternal Twins | Group D: Age 40 - 59 yo Identical Twins | Group E: Age 40 - 59 yo Fraternal Twins | Group F: Age 70 - 100 yo Twins
Number analyzed (Participants) | 16 | 14 | 10 | 20 | 14 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 0 to 28 of study participation
Description: Clinical Assessment performed at each visit
Groups:
- Group F: Age 70 - 100 yo Identical Twins: Individual twins to receive Fluzone® (intramuscular) or High-Dose Fluzone® (intramuscular)
  High-Dose Fluzone® (intramuscular): Licensed seasonal High-Dose trivalent inactivated influenza
  Fluzone® (intramuscular): Licensed seasonal trivalent inactivated influenza
Arm/Group | Group A: Age 8-17 yo Identical Twins | Group B: Age 18-30 yo Identical Twins | Group C: Age 18-30 yo Fraternal Twins | Group D: Age 40 - 59 yo Identical Twins | Group E: Age 40 - 59 yo Fraternal Twins | Group F: Age 70 - 100 yo Identical Twins
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14 | 0/10 | 0/20 | 0/14 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14 | 0/10 | 0/20 | 0/14 | 0/8
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14 | 0/10 | 0/20 | 0/14 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No